CLINICAL TRIAL: NCT06058286
Title: An Implementation Trial of Continuous Quality Improvement for Antenatal Syphilis, HIV and Hepatitis B Detection and Treatment in Indonesia
Brief Title: MENJAGA: Continuous Quality Improvement for Antenatal HIV, Syphilis and Hepatitis B Testing in Indonesia
Acronym: MENJAGA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yanri Wijayanti Subronto, MD, PhD, (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other); Kirby Institute (Other Government)
Responsible Party: Sponsor-Investigator, Yanri Wijayanti Subronto, MD, PhD,, Doctor, Gadjah Mada University
Organization: Gadjah Mada University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 000; MR/T038837/1 (Other Grant/Funding Number: Medical Research Council, UK)
Record Dates: First submitted 2023-09-22; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Hiv; Syphilis; Hepatitis B
Keywords: quality improvement; triple elimination; EMTCT; Antenatal care; Indonesia
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Syphilis; Hepatitis B

STUDY DESIGN:
Masking Description: Because of the nature of the intervention, district health officials and healthcare providers will be aware of allocation. Fieldworkers collecting outcome data and women interviewed for the process evaluation will be masked as to allocation. The team analysing the outcome data and interpreting the results will be masked to the study arm until all primary outcome analyses outlined in the statistical analysis plan are completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous quality improvement of antenatal HIV, syphilis and hepatitis B testing (Experimental): Intervention facilities will receive targeted and enhanced support in line with the continuous quality improvement (CQI) approach, over a period of approximately 12 months, to promote implementation of the national guidelines and sustained provision of routine testing for HIV, syphilis and hepatitis B at least once during pregnancy. District-level CQI coaches will provide training in CQI methods to two facility representatives from each of the 20 intervention arm facilities. The CQI coaches will then work with these facility-level 'CQI advocates' to implement a process of quality improvement to identify and address barriers to antenatal testing.
  Interventions: Other: Continuous quality improvement
- Routine antenatal care and testing (No Intervention): In the control clusters, pregnant women will receive the existing standard of antenatal care, including antenatal testing for HIV, syphilis and hepatitis B (usual care).
  Current Indonesian guidelines recommend antenatal screening and treatment for HIV/syphilis/hepatitis B according to clinical protocols (for syphilis this is a single rapid test with no further confirmation of positive tests before commencing treatment using one injection of penicillin at an ANC clinic; for HIV there are three sequential rapid tests with confirmed cases initiating HIV antiretroviral therapy from the closest Care Support and Treatment clinic within the pregnancy period, and for hepatitis B, pregnant women with a reactive hepatitis B serum antigen test will be referred to a hospital for management based on clinical features)

INTERVENTIONS:
Other: Continuous quality improvement — Continuous quality improvement (CQI) is an approach to develop healthcare providers' capacity to improve quality of care processes and improve adherence to clinical guidelines. Key features of CQI include systematic, data-guided activities, designing interventions (or changes to facility processes) with local conditions in mind, and iterative development and testing of interventions. The approach is based on the premise that valuable improvement in organisational processes can be achieved through bottom-up initiatives of stakeholders and providers. It requires a 'team-based' culture of staff working together to collect and use available data to evaluate the effect of local solutions. Facility staff drive the development of solutions to quality of care shortcomings that they feel are best suited to the local context, and CQI works within existing resource constraints so it does not require large long-term investments to sustain improvements.
  Arms: Continuous quality improvement of antenatal HIV, syphilis and hepatitis B testing

SUMMARY:
Elimination of mother-to-child-transmission (EMTCT) of HIV, syphilis and hepatitis B are key priorities in Indonesia, the fourth most populous country in the world. Despite national guidelines and strong antenatal care attendance, coverage of antenatal screening for these diseases among pregnant women remains extremely limited in Indonesia. The Indonesian government is committed to improving the integration of HIV/syphilis/hepatitis B testing and treatment into the antenatal platform but currently lacks comprehensive evidence on interventions to support this. We will evaluate a low-cost and locally driven intervention based on the principles of continuous quality improvement to strengthen antenatal care and promote screening for HIV, syphilis and hepatitis B. Continuous Quality Improvement (CQI), which involves local antenatal care (ANC) teams systematically collecting and reflecting on local data to inform the design and implementation of service delivery, has been effectively used to strengthen ANC in a number of Sub-Saharan African countries but yet to be comprehensively evaluated in ANC services in Indonesia. This approach holds considerable promise for Indonesia, a highly populous and diverse country where a 'one size fits all' approach to the delivery of quality ANC rarely applies.

DETAILED DESCRIPTION:
Using a cluster-randomized design, we will evaluate the effectiveness, cost-effectiveness, acceptability, fidelity and reach of a multi-faceted Continuous Quality Improvement (CQI) intervention to improve antenatal testing and treatment of HIV, syphilis and hepatitis B at primary level healthcare facilities in Indonesia. Under the CQI approach, facility staff drive the development of solutions to quality of care shortcomings that they feel are best suited to the local context, working within existing resource constraints It is expected that through their engagement in the CQI intervention, ANC facilities will be in a stronger position to identify and address barriers to antenatal testing and treatment of HIV/syphilis/hepatitis B while also helping to strengthen the underlying health system. The study will take place in two districts in West Java, Indonesia. Clusters will consist of twenty facilities in each of the two districts (40 facilities total) that will be randomized with a 1:1 allocation ratio to the intervention arm (trained in CQI methods) and the control arm (providing usual care) using a computer-generated randomization schedule stratified by district. Intervention and control arms will be balanced with respect to the following covariates: type of facility (puskesmas -and facility size (number of antenatal care registrations in the previous year). In each district, the study team will train three district-level CQI coaches in quality improvement methods. The CQI coaches, using a train-the-trainer approach, will then train representatives from the 20 intervention arm facilities. Over approximately 12 months, intervention facilities will receive enhanced support in line with the CQI approach to promote implementation of the national guidelines and sustained provision of routine testing for HIV, syphilis and hepatitis B at least once during pregnancy. Facilities randomised to the control arm will continue to provide ANC services and HIV, syphilis and Hepatitis B testing as per the existing standard of care. The primary outcome is the proportion of women tested for HIV,syphilis and hepatitis during their current pregnancy. Current Indonesian guidelines recommend antenatal screening and treatment for HIV/syphilis/hepatitis B according to clinical protocols (for syphilis this is a single rapid test with no further confirmation of positive tests before commencing treatment using one injection of penicillin at an ANC clinic; for HIV there are three sequential rapid tests with confirmed cases initiating HIV antiretroviral therapy from the closest Care Support and Treatment clinic within the pregnancy period, and for hepatitis B, pregnant women with a reactive hepatitis B serum antigen test will be referred to a hospital for management based on clinical features). The overall aim of this study is to eliminate newborn infection with HIV/syphilis/hepatitis B in Indonesia through improved detection and treatment in pregnant women.

ELIGIBILITY:
This is cluster randomized control trial that unit of analysis is health facility. The following are the eligibility criteria for health facilities to be included in the trial:

* Facility with at least 320 first antenatal care visits or registrations per year (based on previous year's data).
* Facility is not currently engaged in another quality improvement intervention or other health-related research.
* Facility expected to provide antenatal care services and HIV/syphilis/hepatitis B testing for the duration of the study.
* Facility recorded 30% or less coverage of HIV testing amongst pregnant women (based on previous year's data).

Exclusion Criteria:

• If any reason is stated by the facility manager for not implementing the intervention if allocated to the intervention arm. Examples of (non-exhaustive) reasons that would exclude the facility are as follows: refusal to participate because of workload concerns or high turnover of staff, etc.

- Facility does not consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of women attending for ANC at one of the participating facilities for the first time, at any point in her pregnancy, who were tested for HIV, syphilis and hepatitis B during that visit. | Over a period of 2-3 months at endline
  This will be calculated as the number of women tested for HIV, syphilis and hepatitis B during their first visit to the facility for antenatal care out of the total number of pregnant women attending the facility for antenatal care for the first time.

SECONDARY OUTCOMES:
Proportion of women tested for HIV during their first visit to the facility for antenatal care | Over a period of 2-3 months at baseline and endline
  This will be calculated as the number of women tested for HIV during their first visit to the facility for antenatal care out of the total number of pregnant women attending the facility for antenatal care for the first time.
Proportion of women tested for syphilis during their first visit to the facility for antenatal care | Over a period of 2-3 months at baseline and endline
  This will be calculated as the number of women tested for syphilis during their first visit to the facility for antenatal care out of the total number of pregnant women attending the facility for antenatal care for the first time.
Proportion of women tested for hepatitis B during their first visit to the facility for antenatal care | Over a period of 2-3 months at baseline and endline
  This will be calculated as the number of women tested for hepatitis B during their first visit to the facility for antenatal care out of the total number of pregnant women attending the facility for antenatal care for the first time.

CONTACTS AND LOCATIONS:
Locations (1):
- Primary Healthcare Centre in Bandung city and Bogor district, Bandung City and Bogor District, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
On project completion, research data will be deposited in the UK Data Archive and LSHTM Research Data Repository. We will only share de-identified study data files.
Supporting Information: Study Protocol
Time Frame: Data in the repositories will be made accessible to other users (outside of the project) at the end of the analysis and publication period (after 24 months of completion of the project).
Access Criteria: Sharing data with researchers outside the project will be permitted under strict data-sharing agreements and/or user registration. As part of the registration/data-sharing agreement process, users must agree to conditions including: 1) restrictions against attempting to identify participants, 2) commitment to securing the data using appropriate technology, 3) destruction of data after analyses are completed, 4) reporting responsibilities, 5) restrictions on redistribution of data, and 6) proper acknowledgement of the data source.